CLINICAL TRIAL: NCT06498323
Title: Intravenous Tenecteplase Versus Alteplase for Acute Ischemic Stroke Treatment on Mobile Stroke Units, a Prospective Multicenter Randomized Controlled Trial
Brief Title: Intravenous TNK vs TPA for AIS Treatment on MSU,a Prospective Multicenter RCT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Yongchai Nilanont, associate professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 376/2565(IRB1)
Record Dates: First submitted 2022-06-13; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Intravenous; Thrombosis; Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Mobile stroke unit; Intravenous Tenecteplase
MeSH Terms: conditions — Thrombosis; Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tenecteplase (Experimental): Intravenous tenecteplase (0.25mg/kg) will be given in acute ischemic stroke patients on mobile stroke units within 4.5 hours according to the eligibility criteria after randomization allocation.
  Interventions: Drug: tenecteplase
- alteplase (Active Comparator): Intravenous alteplase (0.9mg/kg) will be given in acute ischemic stroke patients on mobile stroke units within 4.5 hours according to the eligibility criteria after randomization allocation.
  Interventions: Drug: tenecteplase

INTERVENTIONS:
Drug: tenecteplase — Intravenous thrombolytic agents administration

SUMMARY:
Acute ischemic stroke is one of the devastating diseases that increase hospitalization, disabilities, and deaths worldwide. Current treatment with intravenous thrombolytic agent can help reduce disabilities and improve quality of life. Intravenous Alteplase is proven benefit and now used as the first-line drug for acute ischemic stroke with symptom onset less than 4.5 hours and without contraindications.

Tenecteplase, a genetically engineered tissue-type plasminogen activator, has been questioned to treat acute ischemic stroke instead of intravenous alteplase. Tenecteplase has more advantages over alteplase including higher fibrin specificity, longer half-life and easier to administer as a single intravenous bolus. The efficacy and safety of intravenous tenecteplase has been studied recently. In 2017, A phase 3 randomized open-label, blinded trial (NOR-TEST) 6 showed that there were no significant differences in efficacy and safety between tenecteplase and alteplase in mild stroke patients. A study in 2020, in the setting of acute large artery occlusion, Tenecteplase resulted in a better 90-day neurological outcome and provided more benefits in reperfusion before endovascular thrombectomy10. Regarding safety concerns, tenecteplase showed no significant higher incidence of intracerebral hemorrhage. Administration, tenecteplase might be better in the setting of the case on mobile stroke units. Assuming, earlier reperfusion by thrombolytic drug may have improved patient's neurologic outcomes. We aim to compare the efficacy and safety between intravenous tenecteplase and alteplase in acute ischemic stroke patients given on mobile stroke units within 4.5 hours after symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as Acute ischemic stroke within 4.5 hr of symptom onset
* Age > 18 years old
* No contraindication for thrombolytic drug
* Informed consent from patients

Exclusion Criteria:

* Diagnosed as Acute ischemic stroke with more than 4.5 hours of symptom onset or uncontained onset
* Have contraindication for thrombolytic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
mRS Score | at 3 months
  mRS Score

SECONDARY OUTCOMES:
NIHSS Score at 24 hrs | at 24 hours
  NIHSS Score at 24 hrs after intravenous tenecteplase

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Stroke Center,Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campbell BCV, Mitchell PJ, Churilov L, Yassi N, Kleinig TJ, Dowling RJ, Yan B, Bush SJ, Dewey HM, Thijs V, Scroop R, Simpson M, Brooks M, Asadi H, Wu TY, Shah DG, Wijeratne T, Ang T, Miteff F, Levi CR, Rodrigues E, Zhao H, Salvaris P, Garcia-Esperon C, Bailey P, Rice H, de Villiers L, Brown H, Redmond K, Leggett D, Fink JN, Collecutt W, Wong AA, Muller C, Coulthard A, Mitchell K, Clouston J, Mahady K, Field D, Ma H, Phan TG, Chong W, Chandra RV, Slater LA, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Bladin CF, Sharma G, Desmond PM, Parsons MW, Donnan GA, Davis SM; EXTEND-IA TNK Investigators. Tenecteplase versus Alteplase before Thrombectomy for Ischemic Stroke. N Engl J Med. 2018 Apr 26;378(17):1573-1582. doi: 10.1056/NEJMoa1716405. PMID 29694815
- [Result] Huang X, Cheripelli BK, Lloyd SM, Kalladka D, Moreton FC, Siddiqui A, Ford I, Muir KW. Alteplase versus tenecteplase for thrombolysis after ischaemic stroke (ATTEST): a phase 2, randomised, open-label, blinded endpoint study. Lancet Neurol. 2015 Apr;14(4):368-76. doi: 10.1016/S1474-4422(15)70017-7. Epub 2015 Feb 26. PMID 25726502
- [Result] Haley EC Jr, Thompson JL, Grotta JC, Lyden PD, Hemmen TG, Brown DL, Fanale C, Libman R, Kwiatkowski TG, Llinas RH, Levine SR, Johnston KC, Buchsbaum R, Levy G, Levin B; Tenecteplase in Stroke Investigators. Phase IIB/III trial of tenecteplase in acute ischemic stroke: results of a prematurely terminated randomized clinical trial. Stroke. 2010 Apr;41(4):707-11. doi: 10.1161/STROKEAHA.109.572040. Epub 2010 Feb 25. PMID 20185783
- [Result] Parsons M, Spratt N, Bivard A, Campbell B, Chung K, Miteff F, O'Brien B, Bladin C, McElduff P, Allen C, Bateman G, Donnan G, Davis S, Levi C. A randomized trial of tenecteplase versus alteplase for acute ischemic stroke. N Engl J Med. 2012 Mar 22;366(12):1099-107. doi: 10.1056/NEJMoa1109842. PMID 22435369
- [Result] Logallo N, Novotny V, Assmus J, Kvistad CE, Alteheld L, Ronning OM, Thommessen B, Amthor KF, Ihle-Hansen H, Kurz M, Tobro H, Kaur K, Stankiewicz M, Carlsson M, Morsund A, Idicula T, Aamodt AH, Lund C, Naess H, Waje-Andreassen U, Thomassen L. Tenecteplase versus alteplase for management of acute ischaemic stroke (NOR-TEST): a phase 3, randomised, open-label, blinded endpoint trial. Lancet Neurol. 2017 Oct;16(10):781-788. doi: 10.1016/S1474-4422(17)30253-3. Epub 2017 Aug 2. PMID 28780236
- [Result] Nepal G, Kharel G, Ahamad ST, Basnet B. Tenecteplase versus Alteplase for the Management of Acute Ischemic Stroke in a Low-income Country-Nepal: Cost, Efficacy, and Safety. Cureus. 2018 Feb 9;10(2):e2178. doi: 10.7759/cureus.2178. PMID 29651371
- [Result] Muir KW. Should Tenecteplase Replace Alteplase for Acute Thrombolysis? Stroke. 2021 Mar;52(3):1091-1093. doi: 10.1161/STROKEAHA.120.033593. Epub 2021 Feb 16. No abstract available. PMID 33588587
- [Result] Ronning OM, Logallo N, Thommessen B, Tobro H, Novotny V, Kvistad CE, Aamodt AH, Naess H, Waje-Andreassen U, Thomassen L. Tenecteplase Versus Alteplase Between 3 and 4.5 Hours in Low National Institutes of Health Stroke Scale. Stroke. 2019 Feb;50(2):498-500. doi: 10.1161/STROKEAHA.118.024223. PMID 30602354
- [Result] Katsanos AH, Safouris A, Sarraj A, Magoufis G, Leker RR, Khatri P, Cordonnier C, Leys D, Shoamanesh A, Ahmed N, Alexandrov AV, Tsivgoulis G. Intravenous Thrombolysis With Tenecteplase in Patients With Large Vessel Occlusions: Systematic Review and Meta-Analysis. Stroke. 2021 Jan;52(1):308-312. doi: 10.1161/STROKEAHA.120.030220. Epub 2020 Dec 4. PMID 33272127
- [Result] Hacke W, Kaste M, Bluhmki E, Brozman M, Davalos A, Guidetti D, Larrue V, Lees KR, Medeghri Z, Machnig T, Schneider D, von Kummer R, Wahlgren N, Toni D; ECASS Investigators. Thrombolysis with alteplase 3 to 4.5 hours after acute ischemic stroke. N Engl J Med. 2008 Sep 25;359(13):1317-29. doi: 10.1056/NEJMoa0804656. PMID 18815396